CLINICAL TRIAL: NCT02021318
Title: A Phase 3, Randomized, Open-Label, Active-Controlled Study to Evaluate the Efficacy and Safety of Roxadustat in the Treatment of Anemia in Chronic Kidney Disease Patients Not on Dialysis
Brief Title: Roxadustat in the Treatment of Anemia in Chronic Kidney Disease (CKD) Patients, Not on Dialysis, in Comparison to Darbepoetin Alfa
Acronym: Dolomites
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Collaborators: Kyntra Bio (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1517-CL-0610; 2013-000951-42 (EudraCT Number)
Record Dates: First submitted 2013-12-20; First posted 2013-12-27 (Estimated); Results first posted 2021-03-29 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Anemia in Chronic Kidney Disease in Non-dialysis Patients
Keywords: Non-dialysis; Roxadustat; ASP1517; Chronic Kidney Disease (CKD); Anemia; Hemoglobin
MeSH Terms: conditions — Renal Insufficiency, Chronic; Anemia | interventions — roxadustat; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Roxadustat (Experimental): Participants received roxadustat orally according to the tiered weight-based approach, with starting dose of 70 mg (milligram) given thrice weekly (TIW) to participants weighing up to 70 kg (kilogram) and 100 mg given TIW to participants weighing more than 70 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL (gram per deciliter) and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received roxadustat up to a maximum of 104 weeks.
  Interventions: Drug: Roxadustat
- Darbepoetin alfa (Active Comparator): Participants received initial dose of darbepoetin alfa based upon the weight (either 0.45 μg/kg (microgram per kilogram), as a single subcutaneous or intravenous (IV) injection once weekly or 0.75 μg/kg, as a single subcutaneous injection once every 2 weeks) as per European Summary of Product Characteristics (EU SmPC) along with IV iron supplementation according to the standard of care. Dose-adjustment was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which darbepoetin alfa dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received darbepoetin alfa for up to a maximum of 104 weeks.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Roxadustat — Oral tablet.
  Other Names: ASP1517
  Arms: Roxadustat
Drug: Darbepoetin alfa — Subcutaneous or intravenous injection.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
The primary objective of this study was to evaluate the efficacy of roxadustat compared to darbepoetin alfa in the treatment of anemia in nondialysis-dependent chronic kidney disease (NDD CKD) participants.

DETAILED DESCRIPTION:
This was a phase 3, multicenter, randomized, open-label, active-controlled study. The study was planned to provide key efficacy and safety data for the approval of roxadustat in the treatment of anemia associated with CKD. Participants assigned to roxadustat treatment were administered roxadustat orally as a combination of tablets of different strengths. Participants assigned to darbepoetin alfa treatment were administered darbepoetin alfa subcutaneously or intravenously.

The study consisted of 3 study periods:

* Screening period: up to 6 weeks
* Treatment period: 104 weeks
* Follow-up period: 4 weeks until planned study end (end of year 2)

ELIGIBILITY:
Inclusion Criteria:

* Subject has a diagnosis of CKD, with Kidney Disease Outcomes Quality Initiative (KDOQI) Stage 3, 4 or 5, not on dialysis; with an Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73 m^2 estimated using the abbreviated 4-variable Modification of Diet in Renal Disease (MDRD) equation.
* The mean of the subject's two most recent (prior to randomization) Hb values during the screening period, obtained at least 4 days apart, must be less than or equal to 10.5 g/dL, with a difference of less than or equal to 1.0 g/dL. The last Hb value must be within 10 days prior to randomization.
* Subject is deemed suitable for treatment with Erythropoiesis Stimulating Agent (ESA) using the criteria specified in the Kidney Disease Improving Global Outcomes (KDIGO) 2012 recommendation considering the rate of fall of Hb concentration, prior response to iron therapy, the risk of needing a transfusion, the risks related to ESA therapy and the presence of symptoms attributable to anemia.
* Subject has a serum folate level greater than or equal to lower limit of normal (LLN) at screening.
* Subject has a serum vitamin B12 level greater than or equal to LLN at screening.
* Subject's alanine aminotransferase (ALT) and aspartate aminotransferase (AST) are less than or equal to 3 x upper limit of normal (ULN), and total bilirubin (TBL) is less than or equal to 1.5 x ULN.
* Subject's body weight is 45.0 kg to a maximum of 160.0 kg.
* Male subject must not donate sperm starting from screening, throughout the study period and up to 12 weeks after final study drug administration.

Exclusion Criteria:

* Subject has received any Erythropoiesis Stimulating Agent (ESA) treatment within 12 weeks prior to randomization.
* Subject has received any dose of IV iron within 6 weeks prior to randomization.
* Subject has received a Red Blood Cell (RBC) transfusion within 8 weeks prior to randomization.
* Subject has a known history of myelodysplastic syndrome or multiple myeloma.
* Subject has a known hereditary hematologic disease such as thalassemia or sickle cell anemia, pure red cell aplasia, or other known causes for anemia other than Chronic Kidney Disease (CKD).
* Subject has a known hemosiderosis, hemochromatosis, coagulation disorder, or hypercoagulable condition.
* Subject has a known chronic inflammatory disease that could impact erythropoiesis (e.g., systemic lupus erythematosus, rheumatoid arthritis, celiac disease) even if it is currently in remission.
* Subject is anticipated to undergo elective surgery that is expected to lead to significant blood loss during the study period or anticipated elective coronary revascularization.
* Subject has active or chronic gastrointestinal bleeding.
* Subject has received any prior treatment with roxadustat or a Hypoxia-inducible factor prolyl hydroxylase inhibitor (HIF-PHI).
* Subject has been treated with iron-chelating agents within 4 weeks prior to randomization.
* Subject has a history of chronic liver disease (e.g., cirrhosis or fibrosis of the liver).
* Subject has known New York Heart Association Class III or IV congestive heart failure.
* Subject has had a myocardial infarction, acute coronary syndrome, stroke, seizure, or a thrombotic/thromboembolic event (e.g., deep vein thrombosis or pulmonary embolism) within 12 weeks prior to randomization.
* Subject has one or more contraindications for treatment with darbepoetin alfa:

  * Uncontrolled hypertension, or two or more blood pressure values of SBP greater than or equal to 160 mmHg or DBP greater than or equal to 95 mmHg (within 2 weeks prior to randomization).
  * Known hypersensitivity to darbepoetin alfa, recombinant human erythropoietin, or any of the excipients.
* Subject has a diagnosis or suspicion (e.g., complex kidney cyst of Bosniak Category 2F or higher) of renal cell carcinoma as shown on renal ultrasound within 12 weeks prior to randomization.
* Subject has a history of malignancy, except for the following: cancers determined to be cured or in remission for greater than or equal to 5 years, curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colonic polyps.
* Subject is positive for any of the following:

  * human immunodeficiency virus (HIV).
  * hepatitis B surface antigen (HBsAg).
  * or anti-hepatitis C virus antibody (anti-HCV Ab).
* Subject has an active clinically significant infection that is manifested by White Blood Count (WBC) > Upper Limit of Normal (ULN), and/or fever, in conjunction with clinical signs or symptoms of infection within one week prior to randomization.
* Subject has a known untreated proliferative diabetic retinopathy, diabetic macular edema, macular degeneration or retinal vein occlusion.
* Subject has had any prior organ transplant (that has not been explanted), subject is scheduled for organ transplantation, or subject is likely to initiate renal replacement therapy including dialysis within the first year of the study.
* Subject will be excluded from participation if any of the following apply:

  * subject has received investigational therapy within 30 days or 5 half lives or limit set by national law, whichever is longer, prior to initiation of screening, or
  * any condition which makes the subject unsuitable for study participation.
* Subject has an anticipated use of dapsone in any dose amount or chronic use of acetaminophen/paracetamol >2.0 g/day during the treatment or follow-up period of the study.
* Subject has a history of alcohol or drug abuse within 2 years prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2018-03-23 (Actual); Study Completion 2019-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Europe B.V.
Locations (125):
- Site AT43009, Vienna, Austria
- Belarus (6):
  - Site BY37503, Brest
  - Site BY37501, Grodno
  - Site BY37506, Minsk
  - Site BY37507, Minsk
  - Site BY37505, Minsk
  - Site BY37502, Vitebsk
- Bulgaria (3):
  - Site BG35907, Sofia
  - Site BG35927, Sofia
  - Site BG35916, Varna
- Croatia (5):
  - Site HR38505, Karlovac
  - Site HR38504, Slavonski Brod
  - Site HR38510, Zagreb
  - Site HR38502, Zagreb
  - Site HR38509, Zagreb
- Czechia (3):
  - Site CZ42018, Nový Jičín, CZ
  - Site CZ42008, Liberec
  - Site CZ42021, Prague
- Site FI35810, Helsinki, Finland
- France (6):
  - Site FR33004, Avignon
  - Site FR33009, Colmar
  - Site FR33010, Grenoble
  - Site FR33062, Limoges
  - Site FR33012, Lyon
  - Site FR33007, Saint-Priest-en-Jarez
- Georgia (3):
  - Site GE99503, Tbilisi
  - Site GE99504, Tbilisi
  - Site GE99502, Tbilisi
- Germany (5):
  - Site DE49073, Cloppenburg
  - Site DE49054, Düsseldorf
  - Site DE49065, Hamburg
  - Site DE49075, Heilbronn
  - Site DE49057, Hoyerswerda
- Hungary (5):
  - Site HU36028, Budapest
  - Site HU36029, Budapest
  - Site HU36027, Kistarcsa
  - Site HU36008, Pécs
  - Site HU36046, Velence
- Site IE35301, Cork, Ireland
- Israel (2):
  - Site IL97202, Be’er Ya‘aqov
  - Site IL97215, Haifa
- Latvia (2):
  - Site LV37101, Riga
  - Site LV37104, Ventspils
- Montenegro (2):
  - Site ME38202, Nikšić
  - Site ME38201, Podgorica
- Site NL31005, Utrecht, Netherlands
- North Macedonia (2):
  - Site MK38901, Skopje
  - Site MK38903, Struga
- Poland (7):
  - Site PL48001, Krakow
  - Site PL48066, Puławy
  - Site PL48013, Szczecin
  - Site PL48007, Tarnów
  - Site PL48004, Warsaw
  - Site PL48009, Wroclaw
  - Site PL48059, Zamość
- Portugal (8):
  - Site PT35120, Almada
  - Site PT35131, Braga
  - Site PT35112, Carnaxide
  - Site PT35119, Evora
  - Site PT35118, Lisbon
  - Site PT35133, Matosinhos Municipality
  - Site PT35122, Setúbal
  - Site PT35132, Vila Nova de Gaia
- Romania (4):
  - Site RO40012, Bucharest
  - Site RO40003, Bucharest
  - Site RO40021, Bucharest
  - Site RO40004, Oradea
- Russia (12):
  - Site RU70024, Chelyabinsk
  - Site RU70054, Irkutsk
  - Site RU70047, Moscow
  - Site RU70006, Moscow
  - Site RU70003, Nizhny Novgorod
  - Site RU70004, Omsk
  - Site RU70014, Rostov-on-Don
  - Site RU70011, Saint Petersburg
  - Site RU70002, Saint Petersburg
  - Site RU70060, Saratov
  - Site RU70057, Yaroslavl
  - Site RU70001, Yaroslavl
- Serbia (6):
  - Site RS38102, Belgrade
  - Site RS38105, Belgrade
  - Site RS38103, Belgrade
  - Site RS38104, Belgrade
  - Site RS38117, Kruševac
  - Site RS38101, Niš
- Slovakia (4):
  - Site SK42102, Košice
  - Site SK42109, Košice
  - Site SK42113, Púchov
  - Site SK42116, Senica
- Slovenia (4):
  - Site SI38615, Jesenice
  - Site SI38603, Maribor
  - Site SI38619, Slovenj Gradec
  - Site SI38609, Šempeter pri Gorici
- Spain (9):
  - Site ES34049, Ferrol, A Coruna
  - Site ES34026, Barcelona
  - Site ES34039, Córdoba
  - Site ES34054, Girona
  - Site ES34017, Jaén
  - Site ES34037, Madrid
  - Site ES34010, Madrid
  - Site ES34030, Majadahonda
  - Site ES34041, Santiago de Compostela
- Ukraine (10):
  - Site UA38009, Lviv, Lvivska
  - Site UA38021, Cherkasy
  - Site UA38006, Dnipropetrovsk
  - Site UA38016, Ivano-Frankivsk
  - Site UA38011, Kharkiv
  - Site UA38017, Kiev
  - Site UA38007, Mykolaiv
  - Site UA38008, Odesa
  - Site UA38001, Ternopil
  - Site UA38018, Uzhhorod
- United Kingdom (13):
  - Site GB44098, Dorchester, Dorset
  - Site GB44064, Birmingham
  - Site GB44099, Dartford
  - Site GB44102, Kings Lynn
  - Site GB44081, Leicester
  - Site GB44086, London
  - Site GB44006, London
  - Site GB44082, London
  - Site GB44097, Nottingham
  - Site GB44100, Orpington
  - Site GB44101, Preston
  - Site GB44080, Stoke-on-Trent
  - Site GB44001, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Barratt J, Dellanna F, Portoles J, Choukroun G, De Nicola L, Young J, Dimkovic N, Reusch M. Safety of Roxadustat Versus Erythropoiesis-Stimulating Agents in Patients with Anemia of Non-dialysis-Dependent or Incident-to-Dialysis Chronic Kidney Disease: Pooled Analysis of Four Phase 3 Studies. Adv Ther. 2023 Apr;40(4):1546-1559. doi: 10.1007/s12325-023-02433-0. Epub 2023 Feb 7. PMID 36749544
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=401

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants of ≥ 18 years of age with a diagnosis of chronic kidney disease, with kidney disease outcomes quality initiative stage 3, 4 or 5, anaemic and not receiving dialysis; with an estimated glomerular filtration rate (eGFR) < 60 milliliter per minute per 1.73 meter square (mL/min/1.73 m^2) were enrolled in this study.
Pre-assignment Details: Participants were randomized in a 1:1 ratio to roxadustat or darbepoetin alfa. Randomization was stratified by 4 factors: region, screening hemoglobin (Hb) values (Hb ≤ 8.0 g/dL versus > 8.0 g/dL), history of cardiovascular, cerebrovascular or thromboembolic diseases and screening eGFR (<30 mL/min/1.73 m^2 versus ≥30 mL/min/1.73 m^2 ).
Groups:
- Roxadustat: Participants received roxadustat orally according to the tiered weight-based approach, with starting dose of 70 milligram (mg) given three times weekly (TIW) to participants weighing between 45 kilogram (kg) up to 70 kg and 100 mg given TIW to participants weighing more than 70 kg up to 160 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received roxadustat for up to a maximum of 104 weeks.
- Darbepoetin Alfa: Participants received initial dose of darbepoetin alfa based upon the weight (either 0.45 microgram per kilogram [μg/kg] of body weight, as a single subcutaneous or intravenous [IV] injection once weekly or 0.75 μg/kg of body weight, as a single subcutaneous injection once every 2 weeks) as per European Summary of Product Characteristics (EU SmPC) along with IV iron supplementation according to the standard of care. Dose-adjustment was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 grams per deciliter (g/dL) and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which darbepoetin alfa dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received darbepoetin alfa for up to a maximum of 104 weeks.
Period: Overall Study
Arm/Group | Roxadustat | Darbepoetin Alfa
Started | 323 | 293
Completed | 250 | 230
Not Completed | 73 | 63
Not completed — Adverse Event | 2 | 1
Not completed — Death | 33 | 34
Not completed — Lost to Follow-up | 3 | 3
Not completed — Progressive Disease | 0 | 1
Not completed — Withdrawal by Subject | 30 | 18
Not completed — Physician Decision | 3 | 3
Not completed — Miscellaneous | 2 | 3

BASELINE CHARACTERISTICS:
Population: The analysis population was the safety analysis set which consisted of all randomized participants who received at least one dose of study drug.
Groups:
- Roxadustat: Participants received roxadustat orally according to the tiered weight-based approach, with starting dose of 70 mg given TIW to participants weighing between 45 kg up to 70 kg and 100 mg given TIW to participants weighing more than 70 kg up to 160 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received roxadustat for up to a maximum of 104 weeks.
- Darbepoetin Alfa: Participants received initial dose of darbepoetin alfa based upon the weight (either 0.45 μg/kg of body weight, as a single subcutaneous or IV injection once weekly or 0.75 μg/kg of body weight, as a single subcutaneous injection once every 2 weeks) as per EU SmPC along with IV iron supplementation according to the standard of care. Dose-adjustment was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which darbepoetin alfa dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received darbepoetin alfa for up to a maximum of 104 weeks.
- Total: Total of all reporting groups
Arm/Group | Roxadustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 323 | 293 | 616
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.8 (13.6) | 65.7 (14.4) | 66.3 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 164 | 342
  Male | 145 | 129 | 274
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 9 | 10 | 19
  Race: Black or African American | 8 | 2 | 10
  Race: White | 306 | 281 | 587
Baseline Hb Value [Count of Participants; unit: Participants]
  <=8.0 g/dL | 11 | 10 | 21
  >8.0 g/dL | 312 | 283 | 595

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Hb Response to Treatment at Two Consecutive Visits During the First 24 Weeks of Treatment Without Rescue Therapy
Description: Hb response was measured as Yes or No. Response Yes (responders) was defined as: Hb ≥11.0 g/dL and Hb change from baseline by ≥ 1.0 g/dL, for participants with baseline Hb > 8.0 g/dL; or Hb change from baseline by ≥ 2.0 g/dL, for participants with baseline Hb ≤ 8.0 g/dL at two consecutive visits with available data separated at least 5 days during the first 24 weeks of treatment without having received rescue therapy (red blood cell [RBC] transfusion for all participants or darbepoetin for roxadustat treated participant).
Time Frame: Baseline to week 24
Population: The analysis population was the Per Protocol Set (PPS) which consisted of all Full Analysis Set (FAS) participants who did not meet any of exclusion criteria from the PPS. The FAS consisted of all randomized participants who received at least one dose of study drug and had at least one post-dose valid Hb assessment.
Measure: Number; unit: Percentage of Participants
Groups:
- Roxadustat: Participants received roxadustat orally according to the tiered weight-based approach, with starting dose of 70 mg given TIW to participants weighing between 45 kg up to 70 kg and 100 mg given TIW to participants weighing more than 70 kg up to 160 kg. Dose-titration was performed based upon regular measurement of Hb levels until participants achieved central Hb value of >= 11.0 g/dL and Hb increase from baseline of >= 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which roxadustat dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received roxadustat for up to a maximum of 104 weeks.
- Darbepoetin Alfa: Participants received initial dose of darbepoetin alfa based upon the weight (either 0.45 mcg/kg of body weight, as a single subcutaneous or IV injection once weekly or 0.75 mcg/kg of body weight, as a single subcutaneous injection once every 2 weeks) as per EU SmPC along with IV iron supplementation according to the standard of care. Dose-adjustment was performed based upon regular measurement of Hb levels until participants achieved central Hb value of >= 11.0 g/dL and Hb increase from baseline of >= 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which darbepoetin alfa dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received darbepoetin alfa for up to a maximum of 104 weeks.
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 286 | 273
Percentage of Participants | 89.5 | 78.0
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; A generalized linear model as an approximation for the Miettinen and Nurminen method, adjusted for stratification factors (actual) was used to estimate the difference of proportions and 95% confidence interval; Test type: Non-Inferiority — Non-inferiority of roxadustat versus darbepoetin alfa, margin = -15% (non-inferiority is concluded if the lower limit of the 95% confidence interval of the difference was >-15%); Difference in percentage = 11.51, 95% CI 2-sided [5.66 to 17.36]

2. Secondary Outcome: Change From Baseline in Hb to the Average Hb of Weeks 28 to 36 Without Rescue Therapy Within 6 Weeks Prior to and During This 8-Week Evaluation Period
Description: Baseline Hb was defined as the mean of all available central laboratory Hb values collected before or including the date of first study drug intake (predose).
Time Frame: Baseline and weeks 28 to 36
Population: The analysis population was the PPS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 258 | 249
g/dL | 1.848 (1.079) | 1.839 (0.973)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline Hb, baseline estimated glomerular filtration rate and baseline Hb by visit as continuous covariates; Test type: Non-Inferiority — Non-Inferiority, margin = -0.75 (non-inferiority is concluded if the lower bound of the 95% CI of the least square mean difference (LSM) is > -0.75 g/dL); p = 0.839, Mixed Models Analysis; LSM Difference = 0.015, 95% CI 2-sided [-0.131 to 0.162]

3. Secondary Outcome: Change From Baseline in Low Density Lipoprotein Cholesterol (LDL-C) to the Average LDL-C of Weeks 12 to 28
Description: Baseline LDL-C was defined as the LDL-C value on day 1. If this value was missing, the latest value prior to first study drug administration was used.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 307 | 277
Millimoles per liter (mmol/L) | -0.352 (0.772) | 0.049 (0.705)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline LDL, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = -0.403, 95% CI 2-sided [-0.510 to -0.296]

4. Secondary Outcome: Time to First Intravenous Iron Use
Description: Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to end of treatment (EOT) Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who had received more than one intravenous iron, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Weeks 6, 12, 18, 24, 30 and 36
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Week 6: number analyzed (Participants) | 318 | 280
  Week 6 | 0 [0 to 0] | 2.8 [0.9 to 4.6]
  Week 12: number analyzed (Participants) | 307 | 259
  Week 12 | 1.3 [0 to 2.5] | 6.7 [3.8 to 9.6]
  Week 18: number analyzed (Participants) | 290 | 247
  Week 18 | 3.3 [1.3 to 5.2] | 9.2 [5.8 to 12.6]
  Week 24: number analyzed (Participants) | 281 | 243
  Week 24 | 4.3 [2 to 6.5] | 10.7 [7.1 to 14.3]
  Week 30: number analyzed (Participants) | 272 | 231
  Week 30 | 5.3 [2.8 to 7.8] | 12.6 [8.7 to 16.5]
  Week 36: number analyzed (Participants) | 263 | 226
  Week 36 | 6.7 [3.9 to 9.6] | 13.3 [9.3 to 17.3]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on cardiovascular history and region and adjusting on Hb and eGFR at baseline as continuous covariate. Superiority was declared if the upper bound of the 95% CI was below 1.0; Test type: Superiority; p = 0.004, Regression, Cox; Hazard Ratio (HR) = 0.45, 95% CI 2-sided [0.26 to 0.78]

5. Secondary Outcome: Change From Baseline in Short Form-36 (SF-36) Physical Functioning (PF) Sub-Score to the Average PF Sub Score in Weeks 12 to 28
Description: Baseline SF-36 PF was defined as the SF-36 PF value on Day 1.The SF-36 is a Quality of Life (QoL) instrument designed to assess generic health concepts relevant across age, disease, and treatment groups. The SF-36 contains 36 items that measured eight scales: (1) physical functioning; (2) role limitations due to physical health problems; (3) bodily pain; (4) social functioning; (5) general health perceptions; (6) role limitations due to emotional problems; (7) vitality, energy or fatigue; and (8) mental health. Each scale is transformed into 0-100 score, with higher scores indicating better health status. The SF-36 PF consisted of 11 questions that focused on health and ability to do usual activities, with higher scores indicating better health status.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the PPS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 274 | 256
Units on a scale | 0.913 (7.182) | 2.062 (7.838)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit (weeks 8, 12 and 28) visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline SF-36 PF, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Non-Inferiority — Non-Inferiority, margin = -3 (non-inferiority is concluded if the lower bound of the 95% confidence interval of the LSM difference is > -3 points); p = 0.027, Mixed Models Analysis; LSM Difference = -1.284, 95% CI 2-sided [-2.423 to -0.145]

6. Secondary Outcome: Change From Baseline in SF-36 Vitality (VT) Sub-Score to the Average VT Sub-Score in Weeks 12 to 28
Description: Baseline VT Subscore was defined as the VT value on Day 1. The SF-36 is a QoL instrument designed to assess generic health concepts relevant across age, disease, and treatment groups. The SF-36 vitality has four questions with score range from 0-100 with higher scores indicating better vitality status.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the PPS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 274 | 256
Units on a scale | 4.077 (8.657) | 3.881 (8.76)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit (weeks 8, 12 and 28), visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline SF-36 VT, baseline Hb, baseline eGFR as continuous covariates; Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; p = 0.454, Mixed Models Analysis; LSM Difference = -0.457, 95% CI 2-sided [-1.656 to 0.742]

7. Secondary Outcome: Change From Baseline in Mean Arterial Pressure (MAP) to the Average MAP Value in Weeks 20 to 28: Per Protocol Set
Description: Baseline MAP was defined as the MAP value on Day 1. If this value was missing, the latest value prior to first study drug administration was used. MAP was derived as: MAP = (2/3)*diastolic blood pressure (DBP) + (1/3)*systolic blood pressure (SBP).
Time Frame: Baseline and weeks 20 to 28
Population: The analysis population was the PPS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Groups:
- Darbepoetin Alfa: Participants received initial dose of darbepoetin alfa based upon the weight [either 0.45 mcg/kg of body weight, as a single subcutaneous or IV injection once weekly or 0.75 mcg/kg of body weight, as a single subcutaneous injection once every 2 weeks] as per EU SmPC along with IV iron supplementation according to the standard of care. Dose-adjustment was performed based upon regular measurement of Hb levels until participants achieved central Hb value of >= 11.0 g/dL and Hb increase from baseline of >= 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which darbepoetin alfa dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received darbepoetin alfa for up to a maximum of 104 weeks.
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 265 | 252
Millimeters of mercury (mmHg) | 0.541 (8.549) | 0.588 (8.779)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline MAP, baseline Hb, baseline eGFR as continuous covariates; Test type: Non-Inferiority — Non-Inferiority, margin = 1 mmHg (non-inferiority is concluded if the upper bound of the 95% confidence interval of the LSM difference is < 1); p = 0.547, Mixed Models Analysis; LSM Difference = -0.372, 95% CI 2-sided [-1.587 to 0.842]

8. Secondary Outcome: Time to First Occurrence of Hypertension During Weeks 1 to 36: Per Protocol Set
Description: Hypertension was defined as either SBP ≥ 170 mmHg and an increase from baseline ≥ 20 mmHg or as DBP ≥ 110 mmHg and an increase from baseline ≥ 15 mmHg. For participants who had experienced more than one event, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion. Percentage of participants were reported in this outcome measure.
Time Frame: Weeks 1 to 36
Population: The analysis population was the PPS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 286 | 273
Percentage of Participants | 17.5 | 19.4
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on CV history and Region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Non-Inferiority — Non-inferiority (hazard ratio margin of 1.3). Non-Inferiority was declared if the upper bound of the 95% CI is below 1.3; p = 0.336, Regression, Cox; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.56 to 1.22]

9. Secondary Outcome: Change From Baseline in MAP to the Average MAP Value in Weeks 20 to 28: Full Analysis Set
Description: Baseline MAP was defined as the MAP value on Day 1. If this value was missing, the latest value prior to first study drug administration was used. MAP was derived as: MAP = (2/3)*DBP + (1/3)*SBP.
Time Frame: Baseline and weeks 20 to 28
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 294 | 269
mmHg | 0.635 (8.529) | 0.457 (8.741)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline MAP, baseline Hb, baseline eGFR as continuous covariates; Test type: Superiority; p = 0.818, Mixed Models Analysis; LSM Difference = -0.136, 95% CI 2-sided [-1.299 to 1.026]

10. Secondary Outcome: Time to First Occurrence of Hypertension During Weeks 1 to 36: Full Analysis Set
Description: as for outcome 8
Time Frame: Weeks 1 to 36
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of Participants | 17.4 | 18.8
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on cardiovascular history and region and adjusting on Hb and eGFR at baseline as continuous covariates. Superiority was declared if the upper bound of the 95% CI is lower than 1; Test type: Superiority; p = 0.452, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.60 to 1.26]

11. Secondary Outcome: Change From Baseline in Hb to the Average Hb Value of Weeks 28 to 52 Regardless of Rescue Therapy
Description: Baseline Hb was defined as the mean of all available central laboratory Hb values collected before or including the date of first study drug intake (pre-dose).
Time Frame: Baseline and weeks 28 to 52
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 287 | 266
g/dL | 1.718 (0.958) | 1.673 (0.923)
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.529, Mixed Models Analysis; LSM Difference = 0.038, 95% CI 2-sided [-0.081 to 0.157]

12. Secondary Outcome: Time to First Hb Response During First 24 Weeks of Treatment Regardless of Administration of Rescue Therapy
Description: Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who had experienced more than one event, only their first event was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion. Percentage of participants were reported in this outcome measure.
Time Frame: Weeks 1 to 24
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of Participants | 88.8 | 77.7
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on cardiovascular history and region and adjusting on Hb and eGFR at baseline as continuous covariates; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.64, 95% CI 2-sided [1.38 to 1.96]

13. Secondary Outcome: Time to First Hb Response During First 24 Weeks of Treatment Without Rescue Therapy
Description: as for outcome 12
Time Frame: Weeks 1 to 24
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants | 88.2 | 77.4
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [1.39 to 1.98]

14. Secondary Outcome: Hb Level Averaged Over Weeks 28 to 36, 44 to 52, 72 to 80 and 96 to 104 Without Rescue Therapy
Description: as for outcome 2
Time Frame: Weeks 28 to 36, 44 to 52, 72 to 80 and 96 to 104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
g/dL
  Weeks 28-36: number analyzed (Participants) | 286 | 266
  Weeks 28-36 | 11.403 [11.302 to 11.503] | 11.351 [11.247 to 11.455]
  Weeks 44-52: number analyzed (Participants) | 266 | 251
  Weeks 44-52 | 11.185 [11.082 to 11.289] | 11.188 [11.082 to 11.294]
  Weeks 72-80: number analyzed (Participants) | 241 | 233
  Weeks 72-80 | 11.225 [11.120 to 11.331] | 11.217 [11.110 to 11.324]
  Weeks 96-104: number analyzed (Participants) | 218 | 215
  Weeks 96-104 | 11.102 [10.986 to 11.219] | 11.078 [10.960 to 11.196]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 28-36 - The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline estimated glomerular filtration rate and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.478, Mixed Models Analysis; LSM Difference = 0.051, 95% CI 2-sided [-0.091 to 0.194]
Statistical Analysis 2: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 44-52 - The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline estimated glomerular filtration rate and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.969, Mixed Models Analysis; LSM Difference = -0.003, 95% CI 2-sided [-0.149 to 0.143]
Statistical Analysis 3: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 72-80 - The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline estimated glomerular filtration rate and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.910, Mixed Models Analysis; LSM Difference = 0.009, 95% CI 2-sided [-0.140 to 0.157]
Statistical Analysis 4: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 96-104 - The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline estimated glomerular filtration rate and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.775, Mixed Models Analysis; LSM Difference = 0.024, 95% CI 2-sided [-0.140 to 0.188]

15. Secondary Outcome: Change From Baseline in Hb to Each Postdosing Time Point Regardless Use of Rescue Therapy
Description: as for outcome 11
Time Frame: Baseline and weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 28, 32, 36, 40, 44, 48, 52, 56, 60, 64, 68, 72, 76, 80, 84, 88, 92, 96, 100 and 104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
g/dL
  Hb Change From BL to week 1: number analyzed (Participants) | 308 | 273
  Hb Change From BL to week 1 | 0.381 [0.311 to 0.45] | 0.294 [0.221 to 0.368]
  Hb Change From BL to week 2: number analyzed (Participants) | 314 | 284
  Hb Change From BL to week 2 | 0.862 [0.782 to 0.941] | 0.584 [0.5 to 0.667]
  Hb Change From BL to week 4: number analyzed (Participants) | 311 | 283
  Hb Change From BL to week 4 | 1.508 [1.403 to 1.613] | 1.073 [0.962 to 1.183]
  Hb Change From BL to week 6: number analyzed (Participants) | 306 | 278
  Hb Change From BL to week 6 | 1.845 [1.729 to 1.962] | 1.423 [1.3 to 1.546]
  Hb Change From BL to week 8: number analyzed (Participants) | 301 | 277
  Hb Change From BL to week 8 | 2.063 [1.94 to 2.185] | 1.682 [1.554 to 1.81]
  Hb Change From BL to week 10: number analyzed (Participants) | 301 | 266
  Hb Change From BL to week 10 | 1.941 [1.819 to 2.062] | 1.611 [1.483 to 1.739]
  Hb Change From BL to week 12: number analyzed (Participants) | 288 | 263
  Hb Change From BL to week 12 | 2.33 [2.204 to 2.456] | 2.03 [1.897 to 2.162]
  Hb Change From BL to week 14: number analyzed (Participants) | 293 | 266
  Hb Change From BL to week 14 | 1.904 [1.781 to 2.027] | 1.745 [1.616 to 1.875]
  Hb Change From BL to week 16: number analyzed (Participants) | 289 | 264
  Hb Change From BL to week 16 | 2.177 [2.053 to 2.301] | 1.994 [1.864 to 2.124]
  Hb Change From BL to week 18: number analyzed (Participants) | 286 | 260
  Hb Change From BL to week 18 | 1.783 [1.669 to 1.896] | 1.609 [1.49 to 1.729]
  Hb Change From BL to week 20: number analyzed (Participants) | 282 | 262
  Hb Change From BL to week 20 | 1.986 [1.869 to 2.103] | 1.9 [1.778 to 2.023]
  Hb Change From BL to week 22: number analyzed (Participants) | 276 | 260
  Hb Change From BL to week 22 | 1.584 [1.473 to 1.696] | 1.615 [1.499 to 1.731]
  Hb Change From BL to week 24: number analyzed (Participants) | 283 | 254
  Hb Change From BL to week 24 | 1.493 [1.383 to 1.603] | 1.554 [1.438 to 1.669]
  Hb Change From BL to week 28: number analyzed (Participants) | 276 | 252
  Hb Change From BL to week 28 | 1.803 [1.688 to 1.919] | 1.869 [1.748 to 1.989]
  Hb Change From BL to week 32: number analyzed (Participants) | 269 | 252
  Hb Change From BL to week 32 | 1.687 [1.568 to 1.806] | 1.673 [1.549 to 1.797]
  Hb Change From BL to Week 36: number analyzed (Participants) | 264 | 247
  Hb Change From BL to Week 36 | 1.913 [1.793 to 2.032] | 1.781 [1.657 to 1.905]
  Hb Change From BL to week 40: number analyzed (Participants) | 266 | 254
  Hb Change From BL to week 40 | 1.625 [1.51 to 1.74] | 1.438 [1.32 to 1.556]
  Hb Change From BL to week 44: number analyzed (Participants) | 257 | 248
  Hb Change From BL to week 44 | 1.65 [1.527 to 1.773] | 1.628 [1.502 to 1.754]
  Hb Change From BL to week 48: number analyzed (Participants) | 259 | 245
  Hb Change From BL to week 48 | 1.459 [1.338 to 1.581] | 1.447 [1.322 to 1.572]
  Hb Change From BL to week 52: number analyzed (Participants) | 254 | 242
  Hb Change From BL to week 52 | 1.682 [1.56 to 1.803] | 1.71 [1.585 to 1.835]
  Hb Change From BL to week 56: number analyzed (Participants) | 251 | 243
  Hb Change From BL to week 56 | 1.412 [1.292 to 1.533] | 1.444 [1.321 to 1.567]
  Hb Change From BL to week 60: number analyzed (Participants) | 250 | 242
  Hb Change From BL to week 60 | 1.735 [1.611 to 1.859] | 1.67 [1.543 to 1.796]
  Hb Change From BL to week 64: number analyzed (Participants) | 247 | 236
  Hb Change From BL to week 64 | 1.546 [1.415 to 1.676] | 1.547 [1.414 to 1.681]
  Hb Change From BL to week 68: number analyzed (Participants) | 242 | 229
  Hb Change From BL to week 68 | 1.851 [1.726 to 1.976] | 1.747 [1.62 to 1.875]
  Hb Change From BL to week 72: number analyzed (Participants) | 236 | 227
  Hb Change From BL to week 72 | 1.615 [1.486 to 1.745] | 1.548 [1.416 to 1.68]
  Hb Change From BL to week 76: number analyzed (Participants) | 231 | 225
  Hb Change From BL to week 76 | 1.745 [1.616 to 1.873] | 1.767 [1.636 to 1.898]
  Hb Change From BL to week 80: number analyzed (Participants) | 220 | 220
  Hb Change From BL to week 80 | 1.534 [1.408 to 1.661] | 1.579 [1.451 to 1.707]
  Hb Change From BL to week 84: number analyzed (Participants) | 220 | 219
  Hb Change From BL to week 84 | 1.723 [1.594 to 1.853] | 1.679 [1.548 to 1.809]
  Hb Change From BL to week 88: number analyzed (Participants) | 219 | 220
  Hb Change From BL to week 88 | 1.424 [1.291 to 1.557] | 1.37 [1.236 to 1.504]
  Hb Change From BL to week 92: number analyzed (Participants) | 223 | 215
  Hb Change From BL to week 92 | 1.677 [1.541 to 1.812] | 1.643 [1.505 to 1.78]
  Hb Change From BL to week 96: number analyzed (Participants) | 217 | 213
  Hb Change From BL to week 96 | 1.429 [1.293 to 1.566] | 1.404 [1.266 to 1.542]
  Hb Change From BL to week 100: number analyzed (Participants) | 215 | 204
  Hb Change From BL to week 100 | 1.488 [1.346 to 1.629] | 1.598 [1.454 to 1.742]
  Hb Change From BL to week 104: number analyzed (Participants) | 207 | 201
  Hb Change From BL to week 104 | 1.489 [1.339 to 1.64] | 1.452 [1.299 to 1.606]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Week 1- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.086, Mixed Models Analysis; LSM Difference = 0.087, 95% CI 2-sided [-0.012 to 0.185]
Statistical Analysis 2: Comparison: Roxadustat vs Darbepoetin Alfa; Week 2- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = 0.278, 95% CI 2-sided [0.165 to 0.391]
Statistical Analysis 3: Comparison: Roxadustat vs Darbepoetin Alfa; Week 4- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = 0.435, 95% CI 2-sided [0.284 to 0.586]
Statistical Analysis 4: Comparison: Roxadustat vs Darbepoetin Alfa; Week 6- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = 0.422, 95% CI 2-sided [0.254 to 0.590]
Statistical Analysis 5: Comparison: Roxadustat vs Darbepoetin Alfa; Week 8- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = 0.380, 95% CI 2-sided [0.205 to 0.556]
Statistical Analysis 6: Comparison: Roxadustat vs Darbepoetin Alfa; Week 10- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p < 0.001, Mixed Models Analysis; LSM Difference = 0.330, 95% CI 2-sided [0.155 to 0.505]
Statistical Analysis 7: Comparison: Roxadustat vs Darbepoetin Alfa; Week 12- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.001, Mixed Models Analysis; LSM Difference = 0.300, 95% CI 2-sided [0.119 to 0.482]
Statistical Analysis 8: Comparison: Roxadustat vs Darbepoetin Alfa; Week 14- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.079, Mixed Models Analysis; LSM Difference = 0.159, 95% CI 2-sided [-0.018 to 0.336]
Statistical Analysis 9: Comparison: Roxadustat vs Darbepoetin Alfa; Week 16- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.044, Mixed Models Analysis; LSM Difference = 0.183, 95% CI 2-sided [0.005 to 0.361]
Statistical Analysis 10: Comparison: Roxadustat vs Darbepoetin Alfa; Week 18- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.037, Mixed Models Analysis; LSM Difference = 0.173, 95% CI 2-sided [0.010 to 0.336]
Statistical Analysis 11: Comparison: Roxadustat vs Darbepoetin Alfa; Week 20- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.319, Mixed Models Analysis; LSM Difference = 0.085, 95% CI 2-sided [-0.083 to 0.253]
Statistical Analysis 12: Comparison: Roxadustat vs Darbepoetin Alfa; Week 22- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.709, Mixed Models Analysis; LSM Difference = -0.030, 95% CI 2-sided [-0.190 to 0.129]
Statistical Analysis 13: Comparison: Roxadustat vs Darbepoetin Alfa; Week 24- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.450, Mixed Models Analysis; LSM Difference = -0.061, 95% CI 2-sided [-0.219 to 0.097]
Statistical Analysis 14: Comparison: Roxadustat vs Darbepoetin Alfa; Week 28- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.440, Mixed Models Analysis; LSM Difference = -0.065, 95% CI 2-sided [-0.231 to 0.101]
Statistical Analysis 15: Comparison: Roxadustat vs Darbepoetin Alfa; Week 32- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.874, Mixed Models Analysis; LSM Difference = 0.014, 95% CI 2-sided [-0.157 to 0.184]
Statistical Analysis 16: Comparison: Roxadustat vs Darbepoetin Alfa; Week 36- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.132, Mixed Models Analysis; LSM Difference = 0.131, 95% CI 2-sided [-0.039 to 0.302]
Statistical Analysis 17: Comparison: Roxadustat vs Darbepoetin Alfa; Week 40- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.024, Mixed Models Analysis; LSM Difference = 0.187, 95% CI 2-sided [0.024 to 0.351]
Statistical Analysis 18: Comparison: Roxadustat vs Darbepoetin Alfa; Week 44- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.807, Mixed Models Analysis; LSM Difference = 0.022, 95% CI 2-sided [-0.153 to 0.197]
Statistical Analysis 19: Comparison: Roxadustat vs Darbepoetin Alfa; Week 48- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.890, Mixed Models Analysis; LSM Difference = 0.012, 95% CI 2-sided [-0.160 to 0.185]
Statistical Analysis 20: Comparison: Roxadustat vs Darbepoetin Alfa; Week 52- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.746, Mixed Models Analysis; LSM Difference = -0.029, 95% CI 2-sided [-0.201 to 0.144]
Statistical Analysis 21: Comparison: Roxadustat vs Darbepoetin Alfa; Week 56- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.715, Mixed Models Analysis; LSM Difference = -0.032, 95% CI 2-sided [-0.202 to 0.139]
Statistical Analysis 22: Comparison: Roxadustat vs Darbepoetin Alfa; Week 60- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.463, Mixed Models Analysis; LSM Difference = 0.066, 95% CI 2-sided [-0.110 to 0.242]
Statistical Analysis 23: Comparison: Roxadustat vs Darbepoetin Alfa; Week 64- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.987, Mixed Models Analysis; LSM Difference = -0.002, 95% CI 2-sided [-0.187 to 0.184]
Statistical Analysis 24: Comparison: Roxadustat vs Darbepoetin Alfa; Week 68- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.251, Mixed Models Analysis; LSM Difference = 0.104, 95% CI 2-sided [-0.074 to 0.281]
Statistical Analysis 25: Comparison: Roxadustat vs Darbepoetin Alfa; Week 72- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.473, Mixed Models Analysis; LSM Difference = 0.067, 95% CI 2-sided [-0.117 to 0.251]
Statistical Analysis 26: Comparison: Roxadustat vs Darbepoetin Alfa; Week 76- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.813, Mixed Models Analysis; LSM Difference = -0.022, 95% CI 2-sided [-0.204 to 0.160]
Statistical Analysis 27: Comparison: Roxadustat vs Darbepoetin Alfa; Week 80- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.622, Mixed Models Analysis; LSM Difference = -0.045, 95% CI 2-sided [-0.223 to 0.134]
Statistical Analysis 28: Comparison: Roxadustat vs Darbepoetin Alfa; Week 84- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.632, Mixed Models Analysis; LSM Difference = 0.045, 95% CI 2-sided [-0.138 to 0.227]
Statistical Analysis 29: Comparison: Roxadustat vs Darbepoetin Alfa; Week 88- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.568, Mixed Models Analysis; LSM Difference = 0.055, 95% CI 2-sided [-0.133 to 0.242]
Statistical Analysis 30: Comparison: Roxadustat vs Darbepoetin Alfa; Week 92- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.729, Mixed Models Analysis; LSM Difference = 0.034, 95% CI 2-sided [-0.158 to 0.226]
Statistical Analysis 31: Comparison: Roxadustat vs Darbepoetin Alfa; Week 96- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.797, Mixed Models Analysis; LSM Difference = 0.025, 95% CI 2-sided [-0.168 to 0.218]
Statistical Analysis 32: Comparison: Roxadustat vs Darbepoetin Alfa; Week 100- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.280, Mixed Models Analysis; LSM Difference = -0.110, 95% CI 2-sided [-0.310 to 0.090]
Statistical Analysis 33: Comparison: Roxadustat vs Darbepoetin Alfa; Week 104- The model included treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline Hb, baseline eGFR and baseline Hb by visit as continuous covariates; Test type: Superiority; p = 0.733, Mixed Models Analysis; LSM Difference = 0.037, 95% CI 2-sided [-0.177 to 0.251]

16. Secondary Outcome: Change From Baseline in Hb to Average Hb Value of Weeks 28 to 36, 44 to 52, 72 to 80, 96 to 104 Regardless of Use of Rescue Therapy
Description: as for outcome 2
Time Frame: Baseline and weeks 28 to 36, 44 to 52, 72 to 80 and 96 to 104
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
g/dL
  Hb Change From BL to weeks 28-36: number analyzed (Participants) | 287 | 266
  Hb Change From BL to weeks 28-36 | 1.825 [1.723 to 1.926] | 1.799 [1.694 to 1.905]
  Hb Change From BL to weeks 44-52: number analyzed (Participants) | 267 | 252
  Hb Change From BL to weeks 44-52 | 1.619 [1.513 to 1.724] | 1.62 [1.512 to 1.729]
  Hb Change From BL to weeks 72-80: number analyzed (Participants) | 243 | 233
  Hb Change From BL to weeks 72-80 | 1.652 [1.545 to 1.759] | 1.649 [1.54 to 1.758]
  Hb Change From BL to weeks 96-104: number analyzed (Participants) | 223 | 217
  Hb Change From BL to weeks 96-104 | 1.486 [1.363 to 1.608] | 1.502 [1.378 to 1.626]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.727, Mixed Models Analysis; LSM Difference = 0.026, 95% CI 2-sided [-0.119 to 0.170]
Statistical Analysis 2: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 14, analysis 2]; Test type: Superiority; p = 0.985, Mixed Models Analysis; LSM Difference = -0.001, 95% CI 2-sided [-0.151 to 0.148]
Statistical Analysis 3: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 14, analysis 3]; Test type: Superiority; p = 0.965, Mixed Models Analysis; LSM Difference = 0.003, 95% CI 2-sided [-0.148 to 0.154]
Statistical Analysis 4: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 14, analysis 4]; Test type: Superiority; p = 0.856, Mixed Models Analysis; LSM Difference = -0.016, 95% CI 2-sided [-0.188 to 0.157]

17. Secondary Outcome: Percentage of Hb Values >=10 g/dL and Within 10.0 to 12.0 g/dL in Weeks 28 to 36, 44 to 52, and 96 to 104 Without Use of Rescue Therapy
Description: Percentage for each participant was calculated from the number of Hb values within 10.0-12.0 g/dL / total number of Hb values*100 in weeks 28 to 36, 44 to 52 and 96 to 104 without use of rescue therapy within 6 weeks prior to and during the 8 week evaluation period.
Time Frame: Weeks 28 to 36, 44 to 52 and 96 to 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Percentage of Hb values
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of Hb values
  Weeks 28-36, >= 10: number analyzed (Participants) | 286 | 266
  Weeks 28-36, >= 10 | 93.078 (20.671) | 92.481 (19.876)
  Weeks 28-36, Within 10-12: number analyzed (Participants) | 286 | 266
  Weeks 28-36, Within 10-12 | 67.896 (33.499) | 69.217 (34.171)
  Weeks 44-52, >= 10: number analyzed (Participants) | 266 | 251
  Weeks 44-52, >= 10 | 90.921 (23.123) | 89.416 (24.833)
  Weeks 44-52, Within 10-12: number analyzed (Participants) | 266 | 251
  Weeks 44-52, Within 10-12 | 74.104 (32.119) | 68.931 (35.367)
  Weeks 72-80, >= 10: number analyzed (Participants) | 241 | 233
  Weeks 72-80, >= 10 | 91.494 (20.923) | 90.343 (24.364)
  Weeks 72-80, Within 10-12: number analyzed (Participants) | 241 | 233
  Weeks 72-80, Within 10-12 | 69.71 (32.444) | 67.861 (37.024)
  Weeks 96-104, >= 10: number analyzed (Participants) | 218 | 215
  Weeks 96-104, >= 10 | 90.436 (22.725) | 87.777 (27.03)
  Weeks 96-104, Within 10-12: number analyzed (Participants) | 218 | 215
  Weeks 96-104, Within 10-12 | 72.393 (33.277) | 68.629 (35.352)

18. Secondary Outcome: Time to First Hb Rate of Rise > 2 g/dL Within 4 Weeks
Description: Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who had experienced more than one event, only their first event was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 155 | 188
  Year 0.5 | 45.5 [40 to 51] | 28.9 [23.6 to 34.1]
  Year 1: number analyzed (Participants) | 131 | 171
  Year 1 | 48.8 [43.2 to 54.4] | 30.9 [25.4 to 36.3]
  Year 1.5: number analyzed (Participants) | 104 | 145
  Year 1.5 | 53.4 [47.7 to 59.1] | 35 [29.3 to 40.7]
  Year 2: number analyzed (Participants) | 10 | 22
  Year 2 | 55.3 [49.5 to 61] | 37.8 [31.9 to 43.7]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 1.74, 95% CI 2-sided [1.36 to 2.22]

19. Secondary Outcome: Number of Hospitalizations
Description: The number of hospitalizations per participant were calculated during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Baseline to EOT (up to week 104)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Hospitalizations
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Hospitalizations | 1.5 (2.4) | 1.4 (2.3)

20. Secondary Outcome: Number of Days of Hospitalization Per Year
Description: The number of days of hospitalization per year was calculated as the sum of the durations of all hospitalizations in days (minimum [date of discharge, end of efficacy of emergent period] - date of admission + 1) / (duration of efficacy emergent period in days / 365.25). The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Baseline to EOT (up to week 104)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Days per year
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Days per year | 12.6 (22) | 11.3 (27.7)

21. Secondary Outcome: Time to First Hospitalization
Description: Time to first hospitalization in years was defined in years as: (first event date during the efficacy emergent period - analysis date of first dose intake +1)/365.25, and the 'first event date' was defined as 'date of first admission and 'analysis date of first dose intake. Date of end of efficacy emergent period was defined as as the treatment period up to the EOT visit. For participants who have experienced more than one hospitalization, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 207 | 216
  Year 0.5 | 31.7 [26.5 to 36.8] | 21.8 [17 to 26.7]
  Year 1: number analyzed (Participants) | 162 | 158
  Year 1 | 43.7 [38.2 to 49.3] | 40.4 [34.6 to 46.2]
  Year 1.5: number analyzed (Participants) | 122 | 124
  Year 1.5 | 55.2 [49.6 to 60.9] | 50.2 [44.2 to 56.1]
  Year 2: number analyzed (Participants) | 15 | 24
  Year 2 | 62.3 [56.7 to 67.9] | 56.7 [50.7 to 62.7]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard ratio was calculated using stratified Cox Proportional Hazards regression stratifying on CV history and Region and adjusting on Hb and eGFR at baseline as continuous covariates. Superiority was declared if the upper bound of the 95% CI is below 1.0; Test type: Superiority; p = 0.079, Regression, Cox; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [0.98 to 1.50]

22. Secondary Outcome: Time to First Use of RBC Transfusion
Description: Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who had experienced more than one RBC transfusion, only their first event was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 281 | 263
  Year 0.5 | 3 [1.1 to 4.9] | 2.1 [0.4 to 3.8]
  Year 1: number analyzed (Participants) | 244 | 233
  Year 1 | 7.3 [4.3 to 10.3] | 6.5 [3.5 to 9.5]
  Year 1.5: number analyzed (Participants) | 214 | 207
  Year 1.5 | 10.9 [7.2 to 14.6] | 9.4 [5.8 to 13]
  Year 2: number analyzed (Participants) | 31 | 34
  Year 2 | 13.9 [9.7 to 18.2] | 11.2 [7.3 to 15.1]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.300, Regression, Cox; Hazard Ratio (HR) = 1.30, 95% CI 2-sided [0.79 to 2.11]

23. Secondary Outcome: Number of RBC Packs
Description: The number of RBC packs were calculated as the sum of units transfused during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT visit or last non-missing Hb assessment (for participants who died during the treatment period). Participants with no medication records of RBC have their number of RBC packs set to 0.
Time Frame: Baseline to EOT (up to week 104)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: RBC packs
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
RBC packs | 0.4 (1.20) | 0.4 (1.98)

24. Secondary Outcome: Volume of RBC Transfused
Description: The volume of blood transfused was calculated as the sum of blood volume transfused during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). Participants with no medication records of RBC have their volume set to 0.
Time Frame: Baseline to EOT (up to week 104)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
mL | 97.0 (112.2) | 334.63 (508.40)

25. Secondary Outcome: Number of Particpants Who Received RBC Transfusions
Description: Participants who received RBC transfusions during the efficacy emergent period were reported. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Baseline to EOT (up to week 104)
Population: The analysis population was the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Participants | 38 | 28

26. Secondary Outcome: Time to First Use of Rescue Therapy
Description: Rescue therapy for participants in the roxadustat group included RBC transfusion or ESA therapy and for participants in the darbepoetin alfa group included RBC transfusion only. Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who have experienced more than one use of rescue therapy (i.e. RBC and ESA), only their first event was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 278 | 263
  Year 0.5 | 4 [1.8 to 6.2] | 2.1 [0.4 to 3.8]
  Year 1: number analyzed (Participants) | 241 | 233
  Year 1 | 9.3 [6 to 12.7] | 6.5 [3.5 to 9.5]
  Year 1.5: number analyzed (Participants) | 213 | 207
  Year 1.5 | 13.3 [9.3 to 17.3] | 9.4 [5.8 to 13]
  Year 2: number analyzed (Participants) | 31 | 34
  Year 2 | 16.7 [12.2 to 21.2] | 11.2 [7.3 to 15.1]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 21, analysis 1]; Test type: Superiority; p = 0.055, Regression, Cox; Hazard Ratio (HR) = 1.59, 95% CI 2-sided [0.99 to 2.54]

27. Secondary Outcome: Number of Participants Who Received Rescue Therapy (Composite of RBC Transfusions (All Participants) and Darbepoetin Alfa Use (Roxadustat Treated Participants Only)
Description: Rescue therapy for participants in the roxadustat group included RBC transfusion or ESA therapy and for participants in the darbepoetin alfa group included RBC transfusion only. Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who have experienced more than one use of rescue therapy (i.e. RBC and ESA), only their first event was used.
Time Frame: Baseline to EOT (up to week 104)
Population: The analysis population was the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Participants | 46 | 28

28. Secondary Outcome: Mean Monthly Intravenous Iron Per Participant During Weeks 37 to 52 and 53 to 104
Description: Participants with no or missing medication records of IV Iron had their monthly IV Iron use set to 0 mg.
Time Frame: Weeks 37 to 52 and 53 to 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mg per month
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
mg per month
  Weeks 37 to 52: number analyzed (Participants) | 275 | 258
  Weeks 37 to 52 | 11.028 (64.282) | 13.208 (46.408)
  Weeks 53 to 104: number analyzed (Participants) | 259 | 248
  Weeks 53 to 104 | 18.702 (68.074) | 31.315 (95.306)

29. Secondary Outcome: Time to First Use of IV Iron Supplementation
Description: Participants were analyzed during the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period). For participants who had received more than one IV iron, only their first event following study treatment was used. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 278 | 238
  Year 0.5 | 4.3 [2 to 6.5] | 11.8 [8 to 15.6]
  Year 1: number analyzed (Participants) | 240 | 201
  Year 1 | 10 [6.5 to 13.5] | 19.2 [14.5 to 23.9]
  Year 1.5: number analyzed (Participants) | 206 | 176
  Year 1.5 | 15.9 [11.5 to 20.2] | 24.2 [19 to 29.4]
  Year 2: number analyzed (Participants) | 26 | 30
  Year 2 | 24.9 [18.8 to 31] | 29.1 [23.1 to 35.1]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariate. Superiority was declared if the upper bound of the 95% CI is below 1.0; Test type: Superiority; p = 0.052, Regression, Cox; Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.51 to 1.00]

30. Secondary Outcome: Percentage of Participants With Oral Iron Use Only
Description: Percentage of participants with oral iron use only were calculated based on total number of participants within the efficacy emergent period. The efficacy emergent period was defined as the evaluation period from the analysis date of first dose intake up to EOT Visit or last non-missing Hb assessment (for participants who died during the treatment period).
Time Frame: Day 1 to week 36, weeks 37 to 52, weeks 53 to 104, efficacy emergent period (up to week 104)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of Participants
  During efficacy emergent period | 50.6 | 52.7
  During day 1 to week 36 | 55.3 | 55.1
  During week 37 to 52: number analyzed (Participants) | 275 | 258
  During week 37 to 52 | 55.6 | 55.4
  During week 53 to 104: number analyzed (Participants) | 262 | 249
  During week 53 to 104 | 53.1 | 50.6

31. Secondary Outcome: Change From Baseline to Weeks 8, 28, 52 and 104 in Total Cholesterol
Description: Baseline was defined as the value on Day 1. If baseline value was missing, the latest value prior to first study drug administration was used regardless of fasting.
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
mmol/L
  Change from BL to week 8: number analyzed (Participants) | 311 | 282
  Change from BL to week 8 | -0.92 (0.98) | -0.046 (0.836)
  Change from BL to week 28: number analyzed (Participants) | 285 | 264
  Change from BL to week 28 | -0.531 (1.153) | 0.016 (0.953)
  Change from BL to week 52: number analyzed (Participants) | 256 | 245
  Change from BL to week 52 | -0.524 (1.232) | -0.111 (1.097)
  Change from BL to week 104: number analyzed (Participants) | 215 | 212
  Change from BL to week 104 | -0.695 (1.284) | -0.197 (1.171)

32. Secondary Outcome: Change From Baseline to Weeks 8, 28, 52 and 104 in LDL-C/High-Density Lipoprotein Cholesterol (HDL-C) Ratio
Description: as for outcome 31
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Ratio
  Change from BL to Week 8: number analyzed (Participants) | 310 | 282
  Change from BL to Week 8 | -0.209 (0.665) | -0.049 (0.629)
  Change from BL to Week 28: number analyzed (Participants) | 284 | 262
  Change from BL to Week 28 | 0.016 (0.893) | 0.053 (0.747)
  Change from BL to Week 52: number analyzed (Participants) | 256 | 245
  Change from BL to Week 52 | 0.014 (1.095) | -0.065 (0.871)
  Change from BL to Week 104: number analyzed (Participants) | 215 | 209
  Change from BL to Week 104 | -0.069 (1.579) | 0.012 (1.06)

33. Secondary Outcome: Change From Baseline to Weeks 8, 28, 52 and 104 in Non-HDL Cholesterol
Description: as for outcome 31
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mmoL/L
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
mmoL/L
  Change from BL to week 8: number analyzed (Participants) | 310 | 282
  Change from BL to week 8 | -0.729 (0.9) | -0.045 (0.787)
  Change from BL to week 28: number analyzed (Participants) | 284 | 262
  Change from BL to week 28 | -0.392 (1.098) | 0.02 (0.911)
  Change from BL to week 52: number analyzed (Participants) | 256 | 245
  Change from BL to week 52 | -0.383 (1.19) | -0.114 (1.062)
  Change from BL to week 104: number analyzed (Participants) | 215 | 211
  Change from BL to week 104 | -0.562 (1.162) | -0.15 (1.151)

34. Secondary Outcome: Change From Baseline to Weeks 8, 28, 52 and 104 in Apolipoproteins A1 (ApoA1)
Description: as for outcome 31
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Grams per liter (g/L)
  Change from BL to week 8: number analyzed (Participants) | 310 | 283
  Change from BL to week 8 | -0.184 (0.222) | 0.026 (0.204)
  Change from BL to week 28: number analyzed (Participants) | 287 | 264
  Change from BL to week 28 | -0.104 (0.258) | 0.055 (0.217)
  Change from BL to week 52: number analyzed (Participants) | 254 | 243
  Change from BL to week 52 | -0.12 (0.254) | 0.027 (0.229)
  Change from BL to week 104: number analyzed (Participants) | 214 | 212
  Change from BL to week 104 | -0.116 (0.311) | -0.018 (0.242)

35. Secondary Outcome: Change From Baseline to Weeks 8, 28, 52 and 104 in Apolipoproteins B (ApoB)
Description: as for outcome 31
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Milligrams per deciliter (mg/dL)
  Change from BL to week 8: number analyzed (Participants) | 310 | 283
  Change from BL to week 8 | -16.5 (19.581) | -0.71 (17.791)
  Change from BL to week 28: number analyzed (Participants) | 287 | 264
  Change from BL to week 28 | -10.659 (23.644) | 0.091 (19.672)
  Change from BL to week 52: number analyzed (Participants) | 254 | 243
  Change from BL to week 52 | -10.74 (25.155) | -3.539 (23.811)
  Change from BL to week 104: number analyzed (Participants) | 214 | 212
  Change from BL to week 104 | -13.561 (25.461) | -2.038 (25.857)

36. Secondary Outcome: Change From Baseline to Weeks 8, 28, 52 and 104 in ApoB/ApoA1 Ratio
Description: as for outcome 31
Time Frame: Baseline and weeks 8, 28, 52, 104
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Ratio
  Change from BL to week 8: number analyzed (Participants) | 252 | 252
  Change from BL to week 8 | -0.031 (0.185) | -0.019 (0.13)
  Change from BL to week 28: number analyzed (Participants) | 231 | 234
  Change from BL to week 28 | -0.026 (0.208) | -0.034 (0.159)
  Change from BL to week 52: number analyzed (Participants) | 204 | 217
  Change from BL to week 52 | -0.025 (0.254) | -0.038 (0.191)
  Change from BL to week 104: number analyzed (Participants) | 170 | 187
  Change from BL to week 104 | -0.044 (0.238) | -0.009 (0.218)

37. Secondary Outcome: Number of Participants With Mean LDL Cholesterol < 100 mg/dL
Description: Missing category for fasting only includes non-fasting participants and the participants with missing values.
Time Frame: Weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Participants
  Weeks 12-28: Yes (Regardless Fasting Status) | 147 | 111
  Weeks 12-28: No (Regardless Fasting Status) | 20 | 33
  Weeks 12-28: Missing (Regardless Fasting Status) | 10 | 8
  Weeks 12-28: Yes (Fasting only) | 90 | 69
  Weeks 12-28: No (Fasting only) | 11 | 18
  Weeks 12-28: Missing (Fasting only) | 76 | 65
  Weeks 36-52: Yes (Regardless Fasting Status) | 129 | 104
  Weeks 36-52: No (Regardless Fasting Status) | 26 | 31
  Weeks 36-52: Missing (Regardless Fasting Status) | 22 | 17
  Weeks 36-52: Yes (Fasting only) | 78 | 57
  Weeks 36-52: No (Fasting only) | 15 | 22
  Weeks 36-52: Missing (Fasting only) | 84 | 73

38. Secondary Outcome: Number of Participants Who Had Achieved Antihypertensive Treatment Goal
Description: Achieved antihypertensive treatment goal was defined as SBP < 130 mmHg and DBP < 80 mmHg over an evaluation period defined as the average of available values in weeks 12 to 28 and 36 to 52.
Time Frame: Weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Participants
  Weeks 12-28: Yes | 76 | 64
  Weeks 12-28: No | 228 | 212
  Week 12-28: Missing | 18 | 16
  Weeks 36-52: Yes | 80 | 64
  Weeks 36-52: No | 196 | 193
  Weeks 36-52: Missing | 46 | 35

39. Secondary Outcome: Change From Baseline to the Average of Weeks 12 to 28 and 36 to 52 in SF-36 Physical Component Score (PCS)
Description: Baseline SF-36 PCS was defined as the SF-36 PCS value on day 1.The SF-36 is a QoL instrument designed to assess generic health concepts relevant across age, disease, and treatment groups. The SF-36 contains 36 items that measured eight scales: (1) physical functioning; (2) role limitations due to physical health problems; (3) bodily pain; (4) social functioning; (5) general health perceptions; (6) role limitations due to emotional problems; (7) vitality, energy or fatigue; and (8) mental health. Each scale is transformed into 0-100 score, with higher scores indicating better health status. The PCS was calculated based on all 8 scales and ranged from 5.02-79.78. For each of these above scales, higher scores always indicated better health status.
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Units on a scale
  Change from BL to weeks 12-28: number analyzed (Participants) | 303 | 272
  Change from BL to weeks 12-28 | 1.222 [0.54 to 1.904] | 2.29 [1.576 to 3.004]
  Change from BL to weeks 36-52: number analyzed (Participants) | 271 | 258
  Change from BL to weeks 36-52 | 1.083 [0.358 to 1.808] | 1.686 [0.939 to 2.433]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 12-28 - The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline SF-36 PCS, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p = 0.027, Mixed Models Analysis; LSM Difference = -1.068, 95% CI 2-sided [-2.012 to -0.124]
Statistical Analysis 2: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 36-52 - The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline SF-36 PCS, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p = 0.239, Mixed Models Analysis; LSM Difference = -0.603, 95% CI 2-sided [-1.606 to 0.401]

40. Secondary Outcome: Change From Baseline to the Average of Weeks 12 to 28 and 36 to 52 in Anemia Subscale (AnS) (Additional Concerns) of Functional Assessment of Cancer Therapy-Anemia (FACT-An) Score
Description: Baseline FACT-An AnS was defined as the FACT-An AnS value on day 1. Together with the functional assessment of cancer therapy - general (FACT-G), the AnS is referred to as the FACT-An Total. The AnS scale contains 13 fatigue specific items (the fatigue score) plus 7 items related to anemia. The Anemia AnS score range is 0 to 80. Higher scores indicated better QoL.
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Units on a scale
  Change from BL to weeks 12-28: number analyzed (Participants) | 303 | 272
  Change from BL to weeks 12-28 | 4.71 [3.558 to 5.861] | 5.238 [4.029 to 6.446]
  Change from BL to weeks 36-52: number analyzed (Participants) | 272 | 257
  Change from BL to weeks 36-52 | 3.661 [2.355 to 4.967] | 4.608 [3.252 to 5.964]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 12-28 - The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline FACT-An AnS, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p = 0.517, Mixed Models Analysis; LSM Difference = -0.528, 95% CI 2-sided [-2.127 to 1.072]
Statistical Analysis 2: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 36-52 - The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline FACT-An AnS, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p = 0.308, Mixed Models Analysis; LSM Difference = -0.947, 95% CI 2-sided [-2.771 to 0.877]

41. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 and 36 to 52 in FACT-An Total Score
Description: Baseline FACT-An total score was defined on day 1. Total Fact-An score is composed of FACT-G and Ans scales. FACT-G contains 27 items that cover four dimensions of well-being: physical well being (PWB) - 7 items, functional well being (FWB) - 7 items, social/family well being (SWB) - 7 items, and emotional well being (EWB) - 6 items. The AnS scale contains 13 fatigue specific items (the Fatigue Score) plus 7 items related to anemia. The total score was obtained by summation of the scores from PWB, SWB, EWB, FWB and AnS. The FACT-An Total Score scale range was 0-188. A higher score indicated better QoL.
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Units on a scale
  Change from BL to weeks 12-28: number analyzed (Participants) | 299 | 270
  Change from BL to weeks 12-28 | 7.761 [5.501 to 10.02] | 8.665 [6.299 to 11.031]
  Change from BL to weeks 36-52: number analyzed (Participants) | 268 | 255
  Change from BL to weeks 36-52 | 5.492 [2.915 to 8.069] | 7.259 [4.593 to 9.925]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Week 12-28 - The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline FACT-An total score, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p = 0.570, Mixed Models Analysis; LSM Difference = -0.904, 95% CI 2-sided [-4.032 to 2.224]
Statistical Analysis 2: Comparison: Roxadustat vs Darbepoetin Alfa; Weeks 36-52 -The model included treatment, visit, visit by treatment interaction, region and history of cardiovascular disease as fixed class factors and baseline FACT-An total score, baseline Hb, baseline estimated glomerular filtration rate as continuous covariates; Test type: Superiority; p = 0.334, Mixed Models Analysis; LSM Difference = -1.767, 95% CI 2-sided [-5.354 to 1.820]

42. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 and 36 to 52 in FACT-An Trial Outcome Index (TOI) Score
Description: Baseline FACT-An total TOI Score was defined on day 1. Total FACT-An TOI score is a sum of PWB subscale score, FWB subscale score and Ans scale score. Fact-An TOI scale contains 14 items that cover four dimensions of well-being: PWB -7 items, FWB -7 items, where score range for each PWB subscale and FWB subscale is 0-28. The AnS scale contains 13 fatigue specific items (the Fatigue Score) plus 7 items related to anemia, where score range for Ans scale is 0-80. The total score was obtained by summation of the scores from PWB, FWB and AnS. The FACT-An Total TOI score range was 0-136. A higher score indicated better QoL.
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Units on a scale
  Change from BL to weeks 12-28: number analyzed (Participants) | 300 | 270
  Change from BL to weeks 12-28 | 6.798 (17.830) | 6.876 (16.960)
  Change from BL to weeks 36-52: number analyzed (Participants) | 269 | 255
  Change from BL to weeks 36-52 | 5.602 (19.302) | 5.595 (19.922)

43. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 in Euroqol Questionnaire-5 Dimensions 5 Levels (EQ-5D 5L) Visual Analogue Scale (VAS) Score
Description: Baseline assessment was defined as the value on day 1. The EQ-5D-5L is a self-reported questionnaire, used as a measure of respondents' health related quality of life (HRQoL) and utility values. The EQ-5D consists of the descriptive system and the VAS. The EQ-5D descriptive system comprises 5 dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, extreme problems. The VAS records the respondent's self rated health status on a graduated (0-100) scale, where the endpoints are labeled 'best imaginable health state' and 'worst imaginable health state' with higher scores for higher HRQoL.
Time Frame: Baseline and weeks 12 to 28
Population: The analysis population was the FAS, with participants who had available data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 300 | 271
Units on a scale | 5.137 [3.498 to 6.776] | 4.353 [2.643 to 6.064]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; The model includes treatment, visit, visit by treatment interaction, region and history of CV disease as fixed class factors and baseline EQ-5D 5L VAS, baseline Hb, baseline eGFR as continuous covariates; Test type: Superiority; p = 0.497, Mixed Models Analysis; LSM Difference = 0.784, 95% CI 2-sided [-1.481 to 3.049]

44. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 and 36 to 52 in Work Productivity and Activity Impairment-Anemic Symptoms (WPAI:ANS) Score: Percent Work Time Missed
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to anaemic symptoms; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the anaemic symptoms on productivity while working; Q6=Impact of the anaemic symptoms on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicated greater activity impairment. Multiply scores by 100 to express in percentages. Percent work time missed due to problem: Q2/(Q2+Q4).
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Percent work time
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 35 | 49
Percent work time
  Change from BL to average in weeks 12-28 | -3.793 (32.987) | 0.842 (21)
  Change from BL to average in weeks 36-52: number analyzed (Participants) | 23 | 44
  Change from BL to average in weeks 36-52 | -0.078 (37.047) | 0.216 (23.483)

45. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 and 36 to 52 in WPAI:ANS Score: Percent Impairment While Working
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to anaemic symptoms; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the anaemic symptoms on productivity while working; Q6=Impact of the anaemic symptoms on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicated greater activity impairment. Percent impairment while working due to problem: Q5/10.
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Percent impairment
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 34 | 50
Percent impairment
  Change from BL to weeks 12-28 | -6.618 (22.419) | -2.433 (28.598)
  Change from BL to weeks 36-52: number analyzed (Participants) | 22 | 48
  Change from BL to weeks 36-52 | -7.879 (25.872) | 1.083 (23.102)

46. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 and 36 to 52 in WPAI:ANS Score: Percent Overall Work Impairment
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to anaemic symptoms; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the anaemic symptoms on productivity while working; Q6=Impact of the anaemic symptoms on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicated greater activity impairment. Percent overall work impairment due to problem: Q2/(Q2+Q4)+[(1-(Q2/(Q2+Q4))x(Q5/10)].
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS, with participants who had available data.
Measure: Mean (Standard Deviation); unit: Percent impairment
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 32 | 49
Percent impairment
  Change from BL to weeks 12-28 | -6.112 (23.21) | -1.217 (20.743)
  Change From BL to weeks 36-52: number analyzed (Participants) | 21 | 44
  Change From BL to weeks 36-52 | 2.817 (30.432) | 0.197 (23.431)

47. Secondary Outcome: Change From Baseline to the Average Value of Weeks 12 to 28 and 36 to 52 in WPAI:ANS Score: Percent Activity Impairment
Description: WPAI consisted of 6 questions (Q1=Employment status; Q2=Hours absent from work due to anaemic symptoms; Q3=Hours absent from work due to other reasons; Q4=Hours actually worked; Q5=Impact of the anaemic symptoms on productivity while working; Q6=Impact of the anaemic symptoms on productivity while doing regular daily activities other than work) and a 1-week recall period. Higher WPAI scores indicated greater activity impairment. Percent activity impairment due to problem: Q6/10.
Time Frame: Baseline, weeks 12 to 28 and 36 to 52
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Percent impairment
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percent impairment
  Change from BL to weeks 12-28: number analyzed (Participants) | 300 | 269
  Change from BL to weeks 12-28 | -9.581 (27.367) | -9.34 (27.09)
  Change from BL to weeks 36-52: number analyzed (Participants) | 270 | 254
  Change from BL to weeks 36-52 | -9.365 (28.956) | -8.17 (27.486)

48. Secondary Outcome: Percentage of Participants With Improvements Measured by Patients' Global Impression of Change (PGIC)
Description: The PGIC is a patient-rated instrument that measured change in participant's overall status on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse), when compared to the start of treatment. The percentage of participants presented included very much improved, much improved and minimally improved.
Time Frame: Weeks 8, 12, 28, 52, 76, 104, last assessment (week 108)
Population: The analysis population was the FAS.
Measure: Number; unit: Percentage of Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of Participants
  Week 8 | 76.1 | 79.4
  Week 12 | 83.7 | 83.6
  Week 28 | 83 | 81
  Week 52 | 79.3 | 79.8
  Week 76 | 73 | 74.9
  Week 104 | 71.8 | 76
  Last Assessment | 70.6 | 71.4

49. Secondary Outcome: Change From Baseline to Each Scheduled Measurement in Serum Ferritin
Description: Baseline assessment was assessment from day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104 and end of study (EOS) (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Picomoles per liter (pmol/L)
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Picomoles per liter (pmol/L)
  Week 4: number analyzed (Participants) | 316 | 288
  Week 4 | -190.762 (241.695) | -159.174 (218.981)
  Week 8: number analyzed (Participants) | 307 | 280
  Week 8 | -229.471 (255.677) | -208.356 (309.893)
  Week 12: number analyzed (Participants) | 300 | 271
  Week 12 | -205.722 (271.752) | -201.587 (346.59)
  Week 20: number analyzed (Participants) | 286 | 265
  Week 20 | -99.86 (334.486) | -140.26 (338.512)
  Week 28: number analyzed (Participants) | 286 | 262
  Week 28 | -97.622 (366.153) | -121.574 (348.136)
  Week 36: number analyzed (Participants) | 271 | 256
  Week 36 | -131.801 (355.463) | -120.424 (362.08)
  Week 44: number analyzed (Participants) | 261 | 250
  Week 44 | -120.864 (368.902) | -60.149 (425.455)
  Week 52: number analyzed (Participants) | 254 | 241
  Week 52 | -93.074 (521.433) | -72.383 (459.342)
  Week 60: number analyzed (Participants) | 252 | 243
  Week 60 | -141.264 (355.419) | -47.714 (459.319)
  Week 68: number analyzed (Participants) | 245 | 239
  Week 68 | -110.907 (422.28) | -14.283 (464.714)
  Week 76: number analyzed (Participants) | 235 | 230
  Week 76 | -99.697 (412.982) | 3.424 (615.735)
  Week 84: number analyzed (Participants) | 224 | 221
  Week 84 | -126.615 (403.693) | -1.351 (576.437)
  Week 92: number analyzed (Participants) | 222 | 219
  Week 92 | -98.025 (460.364) | -26.73 (547.371)
  Week 100: number analyzed (Participants) | 216 | 206
  Week 100 | -95.513 (486.758) | 31.391 (750.432)
  Week 104: number analyzed (Participants) | 212 | 208
  Week 104 | -89.276 (476.167) | 26.454 (730.126)
  EOS: number analyzed (Participants) | 245 | 225
  EOS | 78.577 (680.524) | 119.157 (697.39)

50. Secondary Outcome: Change From Baseline to Each Scheduled Measurement in Transferrin Saturation (TSAT)
Description: as for outcome 49
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104 and EOS (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Percentage of saturation
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of saturation
  Week 4: number analyzed (Participants) | 312 | 287
  Week 4 | -6 (10.7) | -2.1 (11.5)
  Week 8: number analyzed (Participants) | 304 | 278
  Week 8 | -5.9 (11.5) | -2.4 (10.6)
  Week 12: number analyzed (Participants) | 294 | 268
  Week 12 | -2.4 (13.2) | -0.5 (12.3)
  Week 20: number analyzed (Participants) | 286 | 263
  Week 20 | 1.6 (13.9) | 2.9 (11.6)
  Week 28: number analyzed (Participants) | 284 | 263
  Week 28 | 1.1 (12.5) | 4 (12.5)
  Week 36: number analyzed (Participants) | 270 | 256
  Week 36 | 1.6 (12) | 3.9 (11.5)
  Week 44: number analyzed (Participants) | 259 | 247
  Week 44 | 0.6 (12) | 4.9 (12.9)
  Week 52: number analyzed (Participants) | 252 | 242
  Week 52 | 1.3 (11.8) | 5.2 (13.2)
  Week 60: number analyzed (Participants) | 250 | 238
  Week 60 | 0.4 (12.4) | 4.8 (12.7)
  Week 68: number analyzed (Participants) | 245 | 237
  Week 68 | 1 (13.4) | 6.3 (13.1)
  Week 76: number analyzed (Participants) | 235 | 228
  Week 76 | 0.1 (12.2) | 6 (13.7)
  Week 84: number analyzed (Participants) | 222 | 220
  Week 84 | 1.1 (12.5) | 6.5 (13.9)
  Week 92: number analyzed (Participants) | 222 | 216
  Week 92 | -0.2 (11.7) | 5.6 (13.8)
  Week 100: number analyzed (Participants) | 214 | 201
  Week 100 | 0.6 (12.4) | 5.8 (14)
  Week 104: number analyzed (Participants) | 210 | 207
  Week 104 | 0.5 (11.9) | 5 (13.3)
  EOS: number analyzed (Participants) | 242 | 222
  EOS | 5.3 (12.3) | 4.7 (13.9)

51. Secondary Outcome: Change From Baseline to Each Scheduled Measurement in Glycated Hemoglobin (HbA1c)
Description: Percentage of change from baseline to each study visit were calculated for HbA1c. Baseline assessment was assessment from Day 1 visit. If baseline value was missing, the value from screening visit was used. In case of missing data, no imputation rules were applied.
Time Frame: Baseline and weeks 12, 28, 36, 44, 60, 84, 104 and EOS (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of HbA1c
  Week 12: number analyzed (Participants) | 296 | 267
  Week 12 | 0.0021 (0.0071) | 0.001 (0.0073)
  Week 28: number analyzed (Participants) | 277 | 256
  Week 28 | 0.0009 (0.0072) | 0.0015 (0.0067)
  Week 36: number analyzed (Participants) | 265 | 252
  Week 36 | 0.0021 (0.0075) | 0.0021 (0.0073)
  Week 44: number analyzed (Participants) | 254 | 249
  Week 44 | 0.0026 (0.0077) | 0.002 (0.0066)
  Week 60: number analyzed (Participants) | 250 | 242
  Week 60 | 0.0025 (0.0083) | 0.0019 (0.0074)
  Week 84: number analyzed (Participants) | 223 | 222
  Week 84 | 0.0024 (0.0093) | 0.0025 (0.0077)
  Week 104: number analyzed (Participants) | 212 | 202
  Week 104 | 0.0018 (0.0086) | 0.002 (0.008)
  EOS: number analyzed (Participants) | 244 | 225
  EOS | 0.0031 (0.0087) | 0.0034 (0.0081)

52. Secondary Outcome: Change From Baseline to Each Scheduled Measurement in Fasting Blood Glucose
Description: as for outcome 49
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104, 106 and EOS (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
mg/dL
  Week 4: number analyzed (Participants) | 169 | 143
  Week 4 | 7 (62.8) | 10.3 (76.9)
  Week 8: number analyzed (Participants) | 168 | 136
  Week 8 | 4.1 (60.1) | 1.3 (40.3)
  Week 12: number analyzed (Participants) | 156 | 134
  Week 12 | 9.3 (64.5) | 7.1 (58.2)
  Week 20: number analyzed (Participants) | 147 | 131
  Week 20 | 6.9 (69.4) | 4.3 (57.9)
  Week 28: number analyzed (Participants) | 137 | 122
  Week 28 | 8.7 (66.9) | 2.8 (37.7)
  Week 36: number analyzed (Participants) | 133 | 126
  Week 36 | 6.4 (52.5) | 3.6 (45.3)
  Week 44: number analyzed (Participants) | 129 | 123
  Week 44 | 3.3 (44.7) | 0.4 (45.1)
  Week 52: number analyzed (Participants) | 129 | 115
  Week 52 | 7.1 (69.7) | 1.1 (41.1)
  Week 60: number analyzed (Participants) | 121 | 104
  Week 60 | 6.6 (65.6) | 6.3 (43.1)
  Week 68: number analyzed (Participants) | 119 | 109
  Week 68 | 3.8 (66.1) | 5.5 (48.2)
  Week 76: number analyzed (Participants) | 113 | 102
  Week 76 | 0.9 (41.9) | 5.8 (55.2)
  Week 84: number analyzed (Participants) | 115 | 101
  Week 84 | 1.4 (49.1) | 12 (57.4)
  Week 92: number analyzed (Participants) | 107 | 95
  Week 92 | 6 (69.5) | 2.1 (46.5)
  Week 100: number analyzed (Participants) | 101 | 87
  Week 100 | 2.7 (45.3) | 4 (48.9)
  Week 104: number analyzed (Participants) | 104 | 90
  Week 104 | -2.6 (60.7) | 1 (48.6)
  Week 106: number analyzed (Participants) | 106 | 92
  Week 106 | -2.4 (31.2) | 9.2 (53.3)
  EOS: number analyzed (Participants) | 116 | 100
  EOS | 2.5 (58.2) | 9.8 (43.6)

53. Secondary Outcome: Change From Baseline to Each Scheduled Measurement in Estimated Glomerular Filtration Rate (eGFR)
Description: as for outcome 49
Time Frame: Baseline and weeks 4, 8, 12, 20, 28, 36, 44, 52, 60, 68, 76, 84, 92, 100, 104, 106 and EOS (up to 108 weeks)
Population: The analysis population was the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Geometric mean ratio
  Week 4: number analyzed (Participants) | 311 | 284
  Week 4 | 1.01 [0.99 to 1.03] | 0.97 [0.95 to 0.99]
  Week 8: number analyzed (Participants) | 300 | 272
  Week 8 | 1.01 [0.98 to 1.03] | 0.96 [0.94 to 0.99]
  Week 12: number analyzed (Participants) | 286 | 261
  Week 12 | 1.02 [1.00 to 1.05] | 0.95 [0.93 to 0.98]
  Week 20: number analyzed (Participants) | 267 | 249
  Week 20 | 0.98 [0.95 to 1.01] | 0.93 [0.90 to 0.96]
  Week 28: number analyzed (Participants) | 252 | 244
  Week 28 | 0.93 [0.89 to 0.96] | 0.89 [0.86 to 0.93]
  Week 36: number analyzed (Participants) | 227 | 227
  Week 36 | 0.93 [0.89 to 0.97] | 0.89 [0.85 to 0.93]
  Week 44: number analyzed (Participants) | 211 | 209
  Week 44 | 0.90 [0.86 to 0.93] | 0.89 [0.84 to 0.93]
  Week 52: number analyzed (Participants) | 200 | 191
  Week 52 | 0.90 [0.86 to 0.94] | 0.88 [0.83 to 0.92]
  Week 60: number analyzed (Participants) | 189 | 182
  Week 60 | 0.90 [0.86 to 0.94] | 0.86 [0.82 to 0.91]
  Week 68: number analyzed (Participants) | 177 | 174
  Week 68 | 0.87 [0.83 to 0.91] | 0.84 [0.79 to 0.89]
  Week 76: number analyzed (Participants) | 167 | 166
  Week 76 | 0.83 [0.78 to 0.88] | 0.84 [0.78 to 0.90]
  Week 84: number analyzed (Participants) | 155 | 157
  Week 84 | 0.83 [0.78 to 0.88] | 0.83 [0.77 to 0.89]
  Week 92: number analyzed (Participants) | 152 | 151
  Week 92 | 0.84 [0.79 to 0.90] | 0.85 [0.79 to 0.90]
  Week 100: number analyzed (Participants) | 145 | 141
  Week 100 | 0.84 [0.78 to 0.89] | 0.86 [0.81 to 0.92]
  Week 104: number analyzed (Participants) | 142 | 140
  Week 104 | 0.84 [0.79 to 0.90] | 0.84 [0.79 to 0.91]
  Week 106: number analyzed (Participants) | 154 | 139
  Week 106 | 0.84 [0.78 to 0.90] | 0.86 [0.79 to 0.92]
  EOS: number analyzed (Participants) | 159 | 146
  EOS | 0.86 [0.81 to 0.91] | 0.85 [0.79 to 0.92]

54. Secondary Outcome: Rate of Progression of Chronic Kidney Disease Measured by eGFR Slope Over Time
Description: Annualized eGFR slope over time was estimated by a random slopes and intercepts model using all available eGFR values (one baseline and all post-treatment values up to EOT period or start of dialysis adjusted on baseline Hb, region, CV history at baseline and the interaction terms (baseline eGFR by timepoint and baseline Hb by timepoint). All assessments collected after initiation of dialysis (acute or chronic) were excluded from the analysis. Baseline assessment was the assessment from day 1 visit. If this value was missing, the value from screening visit was used.
Time Frame: Baseline up to EOS (up to week 108)
Population: The analysis population was the FAS.
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min per 1.73 m^2
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
ml/min per 1.73 m^2 | -2.95 [-3.56 to -2.34] | -2.89 [-3.51 to -2.27]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Test type: Superiority; p = 0.902, Mixed Models Analysis; LSM Difference = -0.05, 95% CI 2-sided [-0.93 to 0.82]

55. Secondary Outcome: Change From Baseline to Each Scheduled Measurement in Urine Albumin/Creatinine Ratio (UACR)
Description: as for outcome 49
Time Frame: Baseline and weeks 12, 24, 36, 52, 64, 76, 88 and 104
Population: The analysis population was the FAS.
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric mean ratio
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Geometric mean ratio
  Week 12: number analyzed (Participants) | 230 | 214
  Week 12 | 1.19 [1.07 to 1.34] | 1.23 [1.1 to 1.38]
  Week 24: number analyzed (Participants) | 225 | 200
  Week 24 | 1.18 [1.06 to 1.33] | 1.22 [1.08 to 1.39]
  Week 36: number analyzed (Participants) | 187 | 181
  Week 36 | 1.22 [1.07 to 1.4] | 1.18 [1.03 to 1.36]
  Week 52: number analyzed (Participants) | 164 | 147
  Week 52 | 1.28 [1.1 to 1.49] | 1.1 [0.92 to 1.32]
  Week 64: number analyzed (Participants) | 149 | 141
  Week 64 | 1.23 [1.03 to 1.46] | 1.11 [0.9 to 1.38]
  Week 76: number analyzed (Participants) | 135 | 133
  Week 76 | 1.39 [1.14 to 1.7] | 1.18 [0.94 to 1.48]
  Week 88: number analyzed (Participants) | 122 | 119
  Week 88 | 1.21 [0.97 to 1.5] | 1.1 [0.86 to 1.39]
  Week 104: number analyzed (Participants) | 109 | 101
  Week 104 | 1.46 [1.17 to 1.82] | 1.18 [0.92 to 1.51]

56. Secondary Outcome: Time to Doubling of Serum Creatinine or Chronic Dialysis or Renal Transplant Compared to Baseline
Description: For participants who had doubled their serum creatinine or had chronic dialysis or renal transplant more than once, only their first occurrence during safety emergent period was used. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of Participants
  Year 0.5: number analyzed (Participants) | 255 | 247
  Year 0.5 | 12.9 [9.1 to 16.6] | 8.6 [5.3 to 11.9]
  Year 1: number analyzed (Participants) | 196 | 186
  Year 1 | 27.4 [22.3 to 32.6] | 27.2 [21.9 to 32.6]
  Year 1.5: number analyzed (Participants) | 155 | 148
  Year 1.5 | 38.2 [32.5 to 44] | 38.8 [32.9 to 44.7]
  Year 2: number analyzed (Participants) | 122 | 113
  Year 2 | 46.5 [40.5 to 52.5] | 45.4 [39.2 to 51.5]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; Hazard Ratio was calculated using stratified Cox Proportional Hazards regression stratifying on CV history and region and adjusting on Hb and eGFR at baseline as continuous covariates. Superiority was declared if the upper bound of the 95% CI was below 1.0; Test type: Superiority; p = 0.960, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.79 to 1.29]

57. Secondary Outcome: Number of Participants With End Stage Renal Disease (ESRD)
Description: Occurrence of end stage renal disease during the study (i.e from day 1 up to the end of study) was defined as at least one of the following: underwent >30 days dialysis therapy, received kidney transplant, planned kidney transplant, physician recommended renal replacement therapy and participant refused therapy, began dialysis and died < 30 days later.
Time Frame: Baseline up to EOS (up to week 108)
Population: The analysis population was the FAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Participants | 110 | 107

58. Secondary Outcome: Time to Chronic Kidney Disease Progression (Composite of Doubling Serum Creatinine, Chronic Dialysis or Renal Transplant, and Death)
Description: Chronic kidney disease progression was defined as date of occurrence of chronic dialysis or date of renal transplant or doubled serum creatinine or date of death, whichever came first. For participants who had chronic dialysis or renal transplant or died, only their first occurrence during the safety emergent period was used. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 255 | 247
  Year 0.5 | 14 [10.1 to 17.9] | 10.2 [6.7 to 13.8]
  Year 1: number analyzed (Participants) | 196 | 186
  Year 1 | 30.9 [25.6 to 36.2] | 29.5 [24.1 to 34.9]
  Year 1.5: number analyzed (Participants) | 155 | 148
  Year 1.5 | 42.1 [36.4 to 47.8] | 42.6 [36.6 to 48.5]
  Year 2: number analyzed (Participants) | 122 | 113
  Year 2 | 49.9 [44 to 55.8] | 51 [44.9 to 57]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p = 0.939, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.79 to 1.25]

59. Secondary Outcome: Time to Chronic Dialysis or Renal Transplant or Death
Description: For participants who had chronic dialysis or renal transplant or died, only their first occurrence during the safety emergent period was used. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments. Data reported was analyzed by Kaplan-Meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula. Percentage of participants were reported in this outcome measure.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 259 | 250
  Year 0.5 | 12.7 [9 to 16.4] | 9.2 [5.8 to 12.6]
  Year 1: number analyzed (Participants) | 207 | 195
  Year 1 | 27.1 [22 to 32.2] | 26.2 [21 to 31.4]
  Year 1.5: number analyzed (Participants) | 169 | 161
  Year 1.5 | 37.1 [31.6 to 42.7] | 37.7 [31.9 to 43.5]
  Year 2: number analyzed (Participants) | 139 | 126
  Year 2 | 42.9 [37.1 to 48.7] | 45.6 [39.6 to 51.7]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p = 0.948, Regression, Cox; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.77 to 1.27]

60. Secondary Outcome: Time to at Least 40% Decrease in eGFR From Baseline, Chronic Dialysis or Renal Transplant
Description: For participants who had at least 40% decrease in eGFR from baseline, chronic dialysis or renal transplant during the safety emergent period, only their first occurrence was used. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments. Data reported was analyzed by kaplan-meier estimate for cumulative proportion and the 95% confidence interval was calculated with Greenwood's formula.
Time Frame: Year 0.5, 1, 1.5 and 2
Population: The analysis population was the FAS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 322 | 292
Percentage of participants
  Year 0.5: number analyzed (Participants) | 248 | 235
  Year 0.5 | 15.4 [11.3 to 19.5] | 13 [9 to 16.9]
  Year 1: number analyzed (Participants) | 178 | 166
  Year 1 | 34.5 [29 to 40] | 35.5 [29.8 to 41.3]
  Year 1.5: number analyzed (Participants) | 133 | 122
  Year 1.5 | 47.2 [41.3 to 53.1] | 50.2 [44.1 to 56.3]
  Year 2: number analyzed (Participants) | 104 | 85
  Year 2 | 55.7 [49.7 to 61.7] | 59.3 [53.2 to 65.3]
Statistical Analysis 1: Comparison: Roxadustat vs Darbepoetin Alfa; [analysis description as in outcome 56, analysis 1]; Test type: Superiority; p = 0.568, Regression, Cox; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.17]

61. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who was given the study drug or who had undergone study procedures and did not necessarily have a causal relationship with this treatment. All AEs collected during the safety emergent period were counted as TEAE. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments. Based on national cancer institute common terminology criteria (NCI-CTCAE), AEs were graded as grade 1=mild, grade 2=moderate, grade 3 =severe or medically significant, grade 4 =life threatening, grade 5 =death related to AE. All reported deaths after the first study drug administration and up to 28 days after the analysis date of last dose were based on last dosing frequency.
Time Frame: From first dose of study drug up to end of study (up to week 108)
Population: The analysis population was the safety analysis set included all randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Roxadustat | Darbepoetin Alfa
Number analyzed (Participants) | 323 | 293
Participants
  TEAE | 296 | 271
  Drug-Related TEAE | 78 | 66
  Serious TEAE | 209 | 181
  Drug-Related Serious TEAE | 18 | 9
  TEAE Leading to Death | 34 | 34
  Drug-Related TEAE Leading to Death | 2 | 0
  TEAE Leading to Withdrawal of Treatment | 25 | 11
  Drug-Related TEAE Leading to Withdraw of Treatment | 7 | 1
  TEAE NCI CTC Grades 3 or Higher | 181 | 164

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to end of study (up to week 108)
Description: Total number of deaths (all causes) includes deaths reported after the time frame above. The safety emergent period was defined as the evaluation period from the analysis date of first drug intake up to 28 days after the end of treatment taking into account the different dosing frequencies of the study treatments.
Groups:
- Darbepoetin Alfa: Participants received initial dose of darbepoetin alfa based upon the weight [either 0.45 μg/kg of body weight, as a single subcutaneous or IV injection once weekly or 0.75 μg/kg of body weight, as a single subcutaneous injection once every 2 weeks] as per EU SmPC along with IV iron supplementation according to the standard of care. Dose-adjustment was performed based upon regular measurement of Hb levels until participants achieved central Hb value of ≥ 11.0 g/dL and Hb increase from baseline of ≥ 1.0 g/dL at two consecutive study visits, separated by at least 5 days. Once target Hb level was reached participants entered maintenance period during which darbepoetin alfa dosage was adjusted every 4 weeks to maintain participants Hb level within the target range of 10.0 g/dL and 12.0 g/dL. Participants received darbepoetin alfa for up to a maximum of 104 weeks.
Arm/Group | Roxadustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 40/323 | 37/293
Serious Adverse Events (participants affected / at risk) | 209/323 | 181/293
Other Adverse Events (participants affected / at risk) | 223/323 | 203/293
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=323) | Darbepoetin Alfa (N=293)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (7)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypocoagulable state (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 3 (3) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 5 (5) | 8 (10)
Angina pectoris (Cardiac disorders) | 0 (0) | 5 (6)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 1 (1)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 2 (2) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 3 (3)
Cardiac failure (Cardiac disorders) | 12 (15) | 10 (15)
Cardiac failure acute (Cardiac disorders) | 3 (3) | 6 (7)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 10 (12)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Long QT syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial fibrosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 1 (1)
Nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 2 (2) | 1 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Trifascicular block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 (1) | 1 (1)
Lown-Ganong-Levine syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Spinocerebellar ataxia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0)
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bloody peritoneal effluent (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis microscopic (Gastrointestinal disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric antral vascular ectasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (3) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oedematous pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (3) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 1 (1)
Reactive gastropathy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 2 (2)
Cardiac death (General disorders) | 2 (2) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 5 (5) | 4 (4)
General physical health deterioration (General disorders) | 1 (1) | 4 (4)
Generalised oedema (General disorders) | 2 (3) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 1 (1) | 1 (1)
Bile duct stone (Hepatobiliary disorders) | 3 (3) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic congestion (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Renal transplant failure (Immune system disorders) | 0 (0) | 1 (1)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 2 (2) | 0 (0)
Acute hepatitis B (Infections and infestations) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial pyelonephritis (Infections and infestations) | 0 (0) | 1 (2)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 3 (3) | 2 (4)
Clostridium colitis (Infections and infestations) | 1 (2) | 1 (3)
Clostridium difficile colitis (Infections and infestations) | 1 (2) | 3 (3)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 3 (4) | 4 (4)
Device related sepsis (Infections and infestations) | 2 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 1 (1) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Gangrene (Infections and infestations) | 4 (4) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Hepatic cyst infection (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 1 (1)
Nosocomial infection (Infections and infestations) | 0 (0) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (2) | 3 (6)
Parotitis (Infections and infestations) | 2 (2) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 3 (3)
Peritonitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 21 (23) | 14 (17)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 1 (2) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 7 (10)
Pyelonephritis chronic (Infections and infestations) | 1 (1) | 0 (0)
Renal cyst infection (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 7 (8) | 9 (9)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 4 (4) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection bacterial (Infections and infestations) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 3 (4)
Urinary tract infection bacterial (Infections and infestations) | 5 (5) | 1 (1)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection pseudomonal (Infections and infestations) | 1 (1) | 1 (1)
Urosepsis (Infections and infestations) | 2 (2) | 3 (3)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arterial bypass occlusion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Arteriovenous fistula site haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 9 (9) | 5 (5)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Shunt malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Shunt occlusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Synovial rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access malfunction (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access site thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 1 (1) | 1 (1)
Blood potassium increased (Investigations) | 2 (2) | 2 (3)
Blood sodium increased (Investigations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 26 (28) | 25 (37)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Occult blood positive (Investigations) | 1 (1) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 7 (10)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Hypervolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 2 (2) | 2 (3)
Mineral deficiency (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (3)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Coma (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (2) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hypoglycaemic coma (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 (1) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 3 (3)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Simple partial seizures (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 6 (6) | 3 (3)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (4) | 3 (3)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 2 (2)
Device dislocation (Product Issues) | 0 (0) | 1 (1)
Device leakage (Product Issues) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 3 (4) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Frustration tolerance decreased (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 7 (8) | 7 (10)
Acute prerenal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Anuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Azotaemia (Renal and urinary disorders) | 1 (1) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
End stage renal disease (Renal and urinary disorders) | 108 (108) | 106 (106)
Haematuria (Renal and urinary disorders) | 1 (2) | 1 (1)
Nephropathy toxic (Renal and urinary disorders) | 1 (1) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal cyst haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal cyst ruptured (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary bladder rupture (Renal and urinary disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bronchopulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Pulmonary vasculitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (3)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Panniculitis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic intramural haematoma (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure fluctuation (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 1 (1)
Embolism arterial (Vascular disorders) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 1 (1) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 8 (11) | 5 (6)
Hypertensive crisis (Vascular disorders) | 5 (5) | 5 (6)
Hypertensive emergency (Vascular disorders) | 1 (1) | 1 (1)
Hypotension (Vascular disorders) | 4 (5) | 2 (2)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1)
Iliac artery occlusion (Vascular disorders) | 1 (2) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 3 (4) | 4 (4)
Peripheral artery occlusion (Vascular disorders) | 1 (1) | 0 (0)
Peripheral artery stenosis (Vascular disorders) | 1 (2) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 4 (6) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.95% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Roxadustat (N=323) | Darbepoetin Alfa (N=293)
Atrial fibrillation (Cardiac disorders) | 16 (18) | 11 (15)
Constipation (Gastrointestinal disorders) | 21 (23) | 15 (18)
Diarrhoea (Gastrointestinal disorders) | 27 (38) | 28 (36)
Nausea (Gastrointestinal disorders) | 35 (40) | 24 (26)
Vomiting (Gastrointestinal disorders) | 21 (31) | 19 (22)
Oedema peripheral (General disorders) | 48 (59) | 36 (52)
Bronchitis (Infections and infestations) | 21 (27) | 17 (21)
Urinary tract infection (Infections and infestations) | 17 (24) | 24 (29)
Viral upper respiratory tract infection (Infections and infestations) | 29 (33) | 25 (30)
Glomerular filtration rate decreased (Investigations) | 33 (35) | 28 (30)
Hyperkalaemia (Metabolism and nutrition disorders) | 34 (38) | 39 (44)
Hyperphosphataemia (Metabolism and nutrition disorders) | 28 (29) | 15 (18)
Iron deficiency (Metabolism and nutrition disorders) | 20 (24) | 24 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 18 (21) | 14 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (22) | 16 (19)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 25 (33) | 15 (20)
Dizziness (Nervous system disorders) | 16 (20) | 13 (15)
Headache (Nervous system disorders) | 20 (23) | 12 (12)
Insomnia (Psychiatric disorders) | 19 (19) | 8 (9)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 12 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (27) | 13 (13)
Hypertension (Vascular disorders) | 93 (129) | 97 (149)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study after Sponsor publication of multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT02021318/Prot_002.pdf
  • Statistical Analysis Plan (2018-09-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT02021318/SAP_003.pdf